CLINICAL TRIAL: NCT03027726
Title: Prevention of Diabetes in Overweight/Obese Preadolescent Children Through a Family-based Intervention Program Including Supervised Exercise; the PREDIKID Study
Brief Title: Prevention of Diabetes in Overweight/Obese Preadolescent Children
Acronym: PREDIKID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); Universidad Pública de Navarra (Other)
Responsible Party: Principal Investigator, IDOIA LABAYEN, Professor, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEP2016-78377-R
Record Dates: First submitted 2017-01-16; First posted 2017-01-23 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Overweight Children With Type 2 Diabetes Risk
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Family-based lifestyle education and psycho-educational program
  Interventions: Behavioral: lifestyle and psycho-educational program
- Exercise group (Experimental): Supervised exercise plus family-based lifestyle education and psycho-educational program
  Interventions: Behavioral: lifestyle and psycho-educational program; Other: Exercise plus lifestyle and psycho-educational program

INTERVENTIONS:
Behavioral: lifestyle and psycho-educational program — The family-based healthy lifestyle education and psychological education program will be followed once every two weeks (11 sessions over 22 weeks) for 90 minutes (45 minutes in the healthy lifestyle education program and 45 minutes in the psycho-educational intervention). The sessions of the healthy lifestyle education and psycho-educational interventions will be developed simultaneously and delivered to both parents (or caregivers) and children, separately. The family-based healthy lifestyle education program will be conducted by experienced nutritionists and the psycho-educational program by experienced psychologists in behavior changes
Other: Exercise plus lifestyle and psycho-educational program — The intervention group will attend the same lifestyle education and psycho-educational program plus the exercise program. The exercise group will do exercise 3 days/week, 90 minutes per session, over a 22-week period. The program will be offered to the families five days per week to choose a total of three days/week. Sessions will be designed and supervised by exercise specialists. The duration of training sessions will be 90 minutes of exercise, including warm-up, moderate to vigorous aerobic activities, and strength exercises
  Arms: Exercise group

SUMMARY:
Background: The global pandemic obesity has led to increased risk for prediabetes and type 2 diabetes (T2D).

Objectives: (i) To evaluate the effect of a 22 weeks multidisciplinary intervention program including exercise on T2D risk in pre-adolescents with high risk to develop T2D, and (ii) To identify the profile of microRNA in circulating exosomes and in blood peripheral mononuclear cells in pre-adolescents with high risk to develop T2D and its response to a multidisciplinary intervention program including exercise.

DETAILED DESCRIPTION:
Background: The global pandemic obesity has led to increased risk for prediabetes and type 2 diabetes (T2D).

Objectives: (i) To evaluate the effect of a 22 weeks multidisciplinary intervention program including exercise on T2D risk in pre-adolescents with high risk to develop T2D, and (ii) To identify the profile of microRNA in circulating exosomes and in blood peripheral mononuclear cells in pre-adolescents with high risk to develop T2D and its response to a multidisciplinary intervention program including exercise.

Design, participants and methods: A total of 84 children with high risk of type 2 diabetes mellitus aged 8-12 years will be included and randomly assigned to control (N=42) or intervention (N=42) groups. The control group will receive a family-based lifestyle education and psycho-educational program (2 days/month), while the intervention group will attend the same lifestyle education and psycho-educational program plus the exercise program (3 days/week). The duration of training sessions will be 90 min of exercise, including warm-up, moderate to vigorous aerobic activities, and strength exercises. The following measurements will be evaluated at baseline prior to randomization and after the intervention: fasting, insulin glucose, and hemoglobin A1c; total and abdominal fat (dual X-ray absorptiometry); pancreatic, hepatic and visceral fat (magnetic resonance imaging); systolic and diastolic blood pressure; fasting leptin, adiponectin, fibroblast growth factor-21, fetuin-A, hs-C-reactive protein, tumor necrosis factor-alfa, interleukin (IL)-1beta and IL-6 and lipid profile; carotid intima-media thickness (ultrasonography), microRNA expression in circulating exosomes and in blood peripheral mononuclear cells (MiSeq-Illumina); functional peak aerobic capacity (cardiopulmonary exercise testing and 20m shuttle run test). Changes in dietary habits (food frequency questionnaire and two non-consecutive 24h recalls), physical activity and sleep (accelerometry); sex, age, socioeconomic status and pubertal status will be used as potential confounders.

Discussion/Conclusions: Early prevention and identification of children with high risk to develop T2D could help to reduce the morbidity and mortality associated with the disease.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese children aged between 8 and 12 years, meeting the international criteria for classification for T2D risk and having at least one parent or caregiver willing to participate in the program sessions will be included

Exclusion Criteria:

* Children with any medical condition that could affect the results of the study or that limits physical activity will be excluded

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | Baseline and at the end of the 22 weeks of intervention
  The Homeostasis model assessment index will be calculated as fasting insulin concentration (microU/mL) x fasting glucose concentration (mmol/L)/22.5.
microRNA expression in circulating exosomes and in blood peripheral mononuclear cells | Baseline and at the end of the 22 weeks of intervention
  The expression of miRNAs will be measured in circulating exosomes and in white blood cells (MiSeq-Ilumina)

SECONDARY OUTCOMES:
Ectopic fat: pancreatic and liver fat accumulation | Baseline and at the end of the 22 weeks of intervention
  Hepatic and pancreatic fat will be measured by magnetic resonance
Total, abdominal and visceral adiposity | Baseline and at the end of the 22 weeks of intervention
  Total and abdominal adiposity will be measured by dual energy X-ray absorptiometry. Visceral adiposity will be measured by magnetic resonance imaging
Anthropometry and blood pressure | Baseline and at the end of the 22 weeks of intervention
  Body mass, height and waist circumference will be measured following standard protocols at least twice until consistent measures will be obtained and thereafter, body mass index (BMI) and waist to height ratio will be calculated. Systolic and diastolic blood pressure measurements will be performed following the recommendations for children using an arm blood pressure oscillometric monitor device
Cardiorespiratory fitness | Baseline and at the end of the 22 weeks of intervention
  Cardiorespiratory fitness will be assessed by two different tests: (i) The 20m shuttle run test in which the equation reported by Léger et al. will be used to estimate the maximum oxygen consumption (VO2max, ml/kg/min) from the 20m shuttle run test scores, and (ii) Direct cardiopulmonary exercise progressive incremental treadmill test using the modified American College of Sports Medicine protocol with respiratory gas analysis to exhaustion
Carotid intima-media thickness | Baseline and at the end of the 22 weeks of intervention
  carotid intima-media thickness will be measured by ultrasound according to international recommendations.
Inflammation and biochemical cardiovascular disease risk factors | Baseline and at the end of the 22 weeks of intervention
  Fasting lipid profile (total-, HDL- and LDL-cholesterol, and triglycerides), glucose, insulin, and hemoglobin A1c, cytokines (e.g. tumor necrosis factor alpha and IL-6) adipokines (e.g leptin and adiponectin), hepatokines (fetuin-A and fibroblast growth factor-21), liver enzymes (alanine aminotransferase, aspartate aminotransferase and gamma-glutamyl transferase), C-reactive protein, thyroid hormones (thyroid stimulating hormone, triiodothyronine and free thyroxine), urea, bilirubin and uric acid

OTHER OUTCOMES:
Confounding variable: puberty stage | Baseline
  The pediatrician will evaluate Tanner staging by direct examination with breast palpation in girls and testicular measurement by orchidometer in boys.
Confounding variable:physical activity and sleep | Baseline and at the end of the 22 weeks of intervention
  Children will wear an activity monitor on the wrist for 7 consecutive days for 24 hours to record physical activity intensity levels and patterns, as well as sleeping habits and participants will also complete a diary log
Confounding variable: dietary habits | Baseline and at the end of the 22 weeks of intervention
  Dietary intake will be evaluated by two non-consecutive 24h recalls within a period of seven days by nutritionists and a validated food frequency questionnaire
Confounding variable: sedentary behaviors | Baseline and at the end of the 22 weeks of intervention
  Sedentary behaviors such as watching television, playing computer games, playing video games or phone games, and surfing the Internet will be self-reported by the children using validated questionnaires
Confounding variable: Socio-demographic variables: | Baseline
  Information about socioeconomic status, demographic characteristics and family medical history of obesity, diabetes, dyslipidemia and hypertension will be collected. Socioeconomic status will be evaluated using The Family Affluence Scale (74) and parental education level and parental occupation. As demographic characteristics date of birth, sex, ethnicity and family structure will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Endocrinology Unit of the University Hospital of Araba (HUA), Vitoria-Gasteiz, Araba, Spain

REFERENCES:
- [Background] Medrano M, Maiz E, Maldonado-Martin S, Arenaza L, Rodriguez-Vigil B, Ortega FB, Ruiz JR, Larrarte E, Diez-Lopez I, Sarasua-Miranda A, Tobalina I, Barrenechea L, Perez-Asenjo J, Kannengiesser S, Manhaes-Savio A, Echaniz O, Labayen I. The effect of a multidisciplinary intervention program on hepatic adiposity in overweight-obese children: protocol of the EFIGRO study. Contemp Clin Trials. 2015 Nov;45(Pt B):346-355. doi: 10.1016/j.cct.2015.09.017. Epub 2015 Sep 25. PMID 26408054
- [Derived] Arenaza L, Medrano M, Amasene M, Rodriguez-Vigil B, Diez I, Grana M, Tobalina I, Maiz E, Arteche E, Larrarte E, Huybrechts I, Davis CL, Ruiz JR, Ortega FB, Margareto J, Labayen I. Prevention of diabetes in overweight/obese children through a family based intervention program including supervised exercise (PREDIKID project): study protocol for a randomized controlled trial. Trials. 2017 Aug 10;18(1):372. doi: 10.1186/s13063-017-2117-y. PMID 28793919